CLINICAL TRIAL: NCT00636207
Title: A Sequential, 3-Part, Double-Blind, Randomized, Placebo-Controlled, Single-Rising-Dose and Rising-Multiple-Dose Study in Healthy Subjects and Mild or Moderate Asthmatic Patients to Evaluate the Safety, Tolerability, and Pharmacokinetics of Inhaled MK-0476
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Inhaled Montelukast (MK-0476) in Participants With Mild or Moderate Asthma (MK-0476-380 AM3)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-380; 2008_516 (Other: Merck Registration ID)
Record Dates: First submitted 2008-03-03; First posted 2008-03-14 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Montelukast 0.1 mg (Experimental): Participants receive Montelukast inhalation powder, 0.1 mg.
  * Part I: Administered as a single dose followed by at least a 3-day washout period.
  Interventions: Drug: Montelukast
- Montelukast 0.3 mg (Experimental): Participants receive Montelukast inhalation powder, 0.3 mg.
  * Part I: Administered as a single dose followed by at least a 3-day washout period.
  Interventions: Drug: Montelukast
- Montelukast 1 mg (Experimental): Participants receive Montelukast inhalation powder, 1 mg.
  * Part I: Administered as a single dose followed by at least a 3-day washout period.
  * Part II: Administered once daily (QD) for 5 days followed by at least a 3-day washout period.
  Interventions: Drug: Montelukast
- Montelukast 3 mg (Experimental): Participants receive Montelukast inhalation powder, 3 mg.
  * Part I: Administered as a single dose followed by at least a 3-day washout period.
  * Part II: Administered QD for 5 days followed by at least a 3-day washout period.
  * Part III: Administered QD for 10 days followed by at least a 7-day washout period.
  Interventions: Drug: Montelukast
- Montelukast 10 mg (Experimental): Participants receive Montelukast inhalation powder, 10 mg.
  * Part I: Administered as a single dose followed by at least a 3-day washout period.
  * Part II: Administered QD for 5 days followed by at least a 3-day washout period.
  * Part III: Administered QD for 10 days followed by at least a 7-day washout period.
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): Participants receive Placebo to Montelukast inhalation powder.
  * Part I: Administered as a single dose followed by at least a 3-day washout period.
  * Part II: Administered QD for 5 days followed by at least a 3-day washout period.
  * Part III: Administered QD for 10 days followed by at least a 7-day washout period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — Montelukast dry powder inhaler, 0.1 mg, 0.3 mg, 1 mg, 3 mg or 10 mg
  Other Names: Montelukast Sodium; MK-0476
  Arms: Montelukast 0.1 mg; Montelukast 0.3 mg; Montelukast 1 mg; Montelukast 10 mg; Montelukast 3 mg
Drug: Placebo — Placebo dry powder inhaler
  Arms: Placebo

SUMMARY:
A study to evaluate the safety, tolerability and pharmacokinetics of inhaled Montelukast (MK-0476) in participants with mild or moderate asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 65
* Must have mild or moderate asthma (Part III only)
* Nonsmoker for at least 6 months

Exclusion Criteria:

* History of stroke, chronic seizures or major neurological disorder
* You are nursing
* Drink more than 3 glasses of alcohol a day
* Have allergy to or not able to tolerate lactose
* Have a history of drug abuse in the last 5 years
* Drink more than 6 beverages containing caffeine a day
* Have had surgery, donated blood or participated in another investigational study in the last 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 study sites located in the United States.
Groups:
- Part I - Montelukast: Part I consisted of 6 periods. Participants were to receive single doses of inhaled Montelukast (0.1 mg, 0.3 mg, 0.3 mg repeat, 1 mg, 3 mg or 10 mg). Each dose was separated by at least a 3-day washout period.
- Part I - Montelukast and Placebo: Part I consisted of 6 periods. Participants were to receive single doses of inhaled Montelukast (0.1 mg, 0.3 mg, 0.3 mg repeat, 1 mg, 3 mg or 10 mg) or Placebo. Each dose was separated by at least a 3-day washout period.
- Part II - Montelukast: Part II consisted of 3 periods. Participants in three serial panels (Panels A, B and C) were to receive once daily (QD) doses of inhaled Montelukast (1 mg, 3 mg or 10 mg) administered for 5 consecutive days. Each panel was separated by at least a 3-day washout period.
- Part II - Placebo: Part II consisted of 3 periods. Participants in three serial panels (Panels A, B and C) were to receive QD doses of inhaled Placebo administered for 5 consecutive days. Each panel was separated by at least a 3-day washout period.
- Part III - Montelukast: Part III consisted of 2 periods. Participants in two serial panels (Panels A and B) were to receive QD doses of inhaled Montelukast (3 mg or 10 mg) administered for 10 consecutive days. Each panel was separated by at least a 7-day washout period.
- Part III - Montelukast and Placebo: Part III consisted of 2 periods. Participants in two serial panels (Panels A and B) were to receive QD doses of inhaled Montelukast (3 mg or 10 mg) or Placebo administered for 10 consecutive days. Each panel was separated by at least a 7-day washout period.
- Part III - Placebo: Part III consisted of 2 periods. Participants in two serial panels (Panels A and B) were to receive QD doses of inhaled or Placebo administered for 10 consecutive days. Each panel was separated by at least a 7-day washout period.
Period: Overall Study
Arm/Group | Part I - Montelukast | Part I - Montelukast and Placebo | Part II - Montelukast | Part II - Placebo | Part III - Montelukast | Part III - Montelukast and Placebo | Part III - Placebo
Started | 1 (One participant discontinued after completing Period 2. Doses in Periods 1 and 2 were Montelukast.) | 8 (One participant withdrew consent after completing all study doses.) | 18 | 6 | 9 (One participant withdrew consent after completing all study doses.) | 1 | 3
Completed | 0 | 7 | 18 | 6 | 8 | 1 | 3
Not Completed | 1 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part I: Part I consisted of 6 periods. Participants were to receive single doses of inhaled Montelukast (0.1 mg, 0.3 mg, 0.3 repeat, 1 mg, 3 mg or 10 mg) or Placebo. Each dose was separated by at least a 3-day washout period.
- Part II: Part II consisted of 3 periods. Participants in three serial panels (Panels A, B and C) were to receive once daily (QD) doses of inhaled Montelukast (1 mg, 3 mg or 10 mg) or Placebo administered for 5 consecutive days. Each panel was separated by at least a 3-day washout period.
- Part III: Part III consisted of 2 periods. Participants in two serial panels (Panels A and B) were to receive QD doses of inhaled Montelukast (3 mg or 10 mg) or Placebo administered for 10 consecutive days. Each panel was separated by at least a 7-day washout period.
- Total: Total of all reporting groups
Arm/Group | Part I | Part II | Part III | Total
Number analyzed (Participants) | 9 | 24 | 13 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (10.45) | 31.0 (12.68) | 36.3 (10.32) | 33.8 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 14 | 6 | 22
  Male | 7 | 10 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced At Least One Adverse Event
Time Frame: Up to 14 days after last dose of study drug
Population: Safety Population: All participants who received at least one dose of study drug
Measure: Number; unit: participants
Groups:
- Montelukast 0.1 mg: Participants receiving Montelukast 0.1 mg inhalation powder
- Montelukast 0.3 mg: Participants receiving Montelukast 0.3 mg inhalation powder
- Montelukast 1 mg: Participants receiving Montelukast 1 mg inhalation powder
- Montelukast 3 mg: Participants receiving Montelukast 3 mg inhalation powder
- Montelukast 10 mg: Participants receiving Montelukast 10 mg inhalation powder
- Placebo: Participants receiving Placebo inhalation powder
Arm/Group | Montelukast 0.1 mg | Montelukast 0.3 mg | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 7 | 7 | 12 | 18 | 19 | 18
participants | 2 | 4 | 6 | 9 | 5 | 6

2. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Time Frame: Up to 7 days after last dose of study drug
Population: Safety Population: All participants who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Montelukast 0.1 mg | Montelukast 0.3 mg | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg | Placebo
Number analyzed (Participants) | 7 | 7 | 12 | 18 | 19 | 18
participants | 0 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Area Under the Curve From 0 to 24 Hours (AUC 0-24hr) of Montelukast - Single Dose
Description: Blood samples for assessment of AUC 0-24hr were drawn predose and then at specified timepoints (up to 24 hours postdose) on Day 1 in Part I.
Time Frame: Up to 24 hours postdose
Population: Per Protocol Population: All participants who complied with the protocol
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Groups:
- Montelukast 0.3 mg Repeat: Participants receiving Montelukast 0.3 mg inhalation powder
Arm/Group | Montelukast 0.1 mg | Montelukast 0.3 mg | Montelukast 0.3 mg Repeat | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg
Number analyzed (Participants) | 7 | 7 | 5 | 6 | 6 | 6
ng/mL*hr | NA (NA) — Plasma level below lower limit of quantitation | NA (NA) — Plasma level below lower limit of quantitation | NA (NA) — Plasma level below lower limit of quantitation | 155 (18.5) | 491 (71) | 1600 (260)

4. Primary Outcome: AUC 0-24hr of Montelukast - Multiple Doses
Description: Blood samples for assessment of AUC 0-24hr were drawn predose and then at specified timepoints (up to 24 hours postdose) on Days 1 and 5 in Part II and on Days 1 and 10 in Part III.
Time Frame: Up to 24 hours postdose
Population: Per Protocol Population: All participants who complied with the protocol
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Groups:
- Montelukast 1 mg: Participants receiving Montelukast 1 mg inhalation powder QD
- Montelukast 3 mg: Participants receiving Montelukast 3 mg inhalation powder QD
- Montelukast 10 mg: Participants receiving Montelukast 10 mg inhalation powder QD
Arm/Group | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL*hr
  Part II Day 1 (n=6) | 132 (43.7) | 403 (115) | 1576 (380)
  Part II Day 5 (n=6) | 214 (76.3) | 576 (148) | 1850 (304)
  Part III Day 1 (n=6) | NA (NA) — Not obtained in Part III | 357 (109) | 1500 (521)
  Part III Day 10 (n=6) | NA (NA) — Not obtained in Part III | 526 (133) | 1880 (530)

5. Primary Outcome: Maximum Plasma Concentration (Cmax) of Montelukast - Single Dose
Description: Blood samples for assessment of Cmax were drawn predose and then at specified timepoints (up to 24 hours postdose) on Day 1 in Part I.
Time Frame: Up to 24 hours postdose
Population: Per Protocol Population: All participants who complied with the protocol
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Montelukast 0.1 mg | Montelukast 0.3 mg | Montelukast 0.3 mg Repeat | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg
Number analyzed (Participants) | 7 | 7 | 5 | 6 | 6 | 6
ng/mL | NA (NA) — Plasma level below lower limit of quantitation | 5.10 (0.977) | 5.24 (0.914) | 18.5 (4.15) | 54.3 (12.7) | 224 (47.3)

6. Primary Outcome: Cmax of Montelukast - Multiple Doses
Description: Blood samples for assessment of Cmax were drawn predose and then at specified timepoints (up to 24 hours postdose) on Days 1 and 5 in Part II and on Days 1 and 10 in Part III.
Time Frame: Up to 24 hours postdose
Population: Per Protocol Population: All participants who complied with the protocol
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Part II Day 1 (n=6) | 13.8 (4.96) | 60 (13.1) | 233 (30.2)
  Part II Day 5 (n=6) | 23.4 (6.5) | 76 (15.3) | 242 (38)
  Part III Day 1 (n=6) | NA (NA) — Not obtained in Part III | 44.3 (16.6) | 184 (66.6)
  Part III Day 10 (n=6) | NA (NA) — Not obtained in Part III | 64.8 (13.0) | 225 (84.7)

7. Primary Outcome: Time to Cmax (Tmax) of Montelukast - Single Dose
Description: Blood samples for assessment of Tmax were drawn predose and then at specified timepoints (up to 24 hours postdose) on Day 1 in Part I.
Time Frame: Up to 24 hours postdose
Population: Per Protocol Population: All participants who complied with the protocol
Measure: Median (Full Range); unit: hours
Arm/Group | Montelukast 0.1 mg | Montelukast 0.3 mg | Montelukast 0.3 mg Repeat | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg
Number analyzed (Participants) | 7 | 7 | 5 | 6 | 6 | 6
hours | NA [NA to NA] — Plasma level below lower limit of quantitation | 2.5 [0.8 to 4.0] | 4.0 [0.5 to 4.0] | 2.4 [0.5 to 7.0] | 0.8 [0.5 to 4.0] | 0.5 [0.5 to 4.0]

8. Primary Outcome: Tmax of Montelukast - Multiple Doses
Description: Blood samples for assessment of Tmax were drawn predose and then at specified timepoints (up to 24 hours postdose) on Days 1 and 5 in Part II and on Days 1 and 10 in Part III.
Time Frame: Up to 24 hours postdose
Population: Per Protocol Population: All participants who complied with the protocol
Measure: Median (Full Range); unit: hours
Arm/Group | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg
Number analyzed (Participants) | 6 | 6 | 6
hours
  Part II Day 1 (n=6) | 2.4 [0.7 to 7] | 0.5 [0.5 to 0.7] | 0.5 [0.5 to 0.7]
  Part II Day 5 (n=6) | 0.7 [0.5 to 0.7] | 0.5 [0.5 to 0.7] | 0.6 [0.5 to 1.0]
  Part III Day 1 (n=6) | NA [NA to NA] — Not obtained in Part III | 0.5 [0.5 to 4.0] | 0.5 [0.2 to 7]
  Part III Day 10 (n=6) | NA [NA to NA] — Not obtained in Part III | 0.5 [0.2 to 0.7] | 0.5 [0.5 to 0.7]

9. Primary Outcome: Apparent Terminal Half Life (t1/2) of Montelukast - Single Dose
Description: Blood samples for assessment of t1/2 were drawn predose and then at specified timepoints (up to 24 hours postdose) on Day 1 in Part I.
Time Frame: Up to 24 hours postdose
Population: Per Protocol Population: All participants who complied with the protocol
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Montelukast 0.1 mg | Montelukast 0.3 mg | Montelukast 0.3 mg Repeat | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg
Number analyzed (Participants) | 7 | 7 | 5 | 6 | 6 | 6
hours | NA (NA) — Plasma level below lower limit of quantitation | NA (NA) — Plasma level below lower limit of quantitation | NA (NA) — Plasma level below lower limit of quantitation | 5.7 (2.1) | 6.9 (0.9) | 5.7 (0.5)

10. Primary Outcome: t1/2 of Montelukast - Multiple Doses
Description: Blood samples for assessment of t1/2 were drawn predose and then at specified timepoints (up to 24 hours postdose) on Days 1 and 5 in Part II and on Days 1 and 10 in Part III.
Time Frame: Up to 24 hours postdose
Population: Per Protocol Population: All participants who complied with the protocol
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg
Number analyzed (Participants) | 6 | 6 | 6
hours
  Part II Day 5 (n=6) | 8.2 (2.5) | 7.6 (2.5) | 7.7 (2.4)
  Part III Day 10 (n=6) | NA (NA) — Not obtained in Part III | 8.1 (1.4) | 7.4 (1.7)

11. Primary Outcome: AUC 0-24hr Accumulation Ratio of Montelukast - Multiple Doses
Description: The AUC 0-24hr Accumulation Ratio of Montelukast was calculated as the geometric mean ratio of AUC 0-24hr on the last day and the first day of a multiple dose regimen: Day 5/Day 1 in Part II and Day 10/Day 1 in Part III.
Time Frame: up to 10 days after first dose of study drug
Population: Per Protocol Population: All participants who complied with the protocol
Measure: Number; unit: ratio
Arm/Group | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg
Number analyzed (Participants) | 6 | 6 | 6
ratio
  Part II (n=6) | 1.61 | 1.44 | 1.2
  Part III (n=6) | NA — Not obtained in Part III | 1.19 | 1.26

12. Primary Outcome: Cmax Accumulation Ratio of Montelukast - Multiple Doses
Description: The Cmax Accumulation Ratio of Montelukast was calculated as the geometric mean ratio of Cmax on the last day and the first day of a multiple dose regimen: Day 5/Day 1 in Part II and Day 10/Day 1 in Part III.
Time Frame: up to 10 days after first dose of study drug
Population: Per Protocol Population: All participants who complied with the protocol
Measure: Number; unit: ratio
Arm/Group | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg
Number analyzed (Participants) | 6 | 6 | 6
ratio
  Part II (n=6) | 1.73 | 1.27 | 1.03
  Part III (n=6) | NA — Not obtained in Part III | 1.03 | 1.22

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose of study drug
Description: Safety Population: All participants who received at least one dose of study drug
Arm/Group | Montelukast 0.1 mg | Montelukast 0.3 mg | Montelukast 1 mg | Montelukast 3 mg | Montelukast 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/12 | 0/18 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 2/7 | 4/7 | 6/12 | 9/18 | 5/19 | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast 0.1 mg (N=7) | Montelukast 0.3 mg (N=7) | Montelukast 1 mg (N=12) | Montelukast 3 mg (N=18) | Montelukast 10 mg (N=19) | Placebo (N=18)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Herpes Simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 5 | 3 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 3 | 2 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Periorbital Oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.